CLINICAL TRIAL: NCT04529044
Title: A Phase II Pilot Study of (Lutetium (177Lu)-DOTATATE in Patients With Metastatic Breast Cancer
Brief Title: 177Lu-DOTATATE for the Treatment of Stage IV or Recurrent Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Advanced Accelerator Applications (Industry); Oregon Health and Science University (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Rodney Pommier, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019489; NCI-2020-04795 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00019489 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Specimen Handling; Ga(III)-DOTATOC; gallium Ga 68 dotatate; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (177Lu-DOTATATE) (Experimental): Patients receive 177Lu-DOTATATE IV over 30-40 minutes during weeks 1, 8, 16, and 24 in the absence of disease progression or unacceptable toxicity. Patients also receive Ga 68-DOTATATE and undergo PET/CT during screening, biopsy as clinically-indicated as well as CT and/or MRI and collection of blood samples throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Gallium Ga 68-DOTATATE; Drug: Lutetium Lu 177 Dotatate; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Radiation: Gallium Ga 68-DOTATATE — Receive 68Ga
  Other Names: (68)Ga-DOTA-TATE; 68Ga-DOTA-0-Tyr3-Octreotate; 68Ga-DOTATATE; Gallium Ga 68 Oxodotreotide; Gallium Oxodotreotide Ga-68; Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial investigates how well 177Lu-DOTATATE works in treating patients with breast cancer that is stage IV or has come back (recurrent). 177Lu-DOTATATE may shrink or destroy the tumor or circulating breast cancer stem cells if they show evidence of the SSTR2. 177Lu-DOTATATE is a targeted therapy that uses DOTATATE, linked to a radioactive agent called 177Lu. DOTATATE attaches to tumor cells with SSTR2 and delivers 177Lu to kill them. Giving 177Lu-DOTATATE may help decrease the number and size of tumors and the number of circulating cancer stem cells in patient's blood for the treatment of patients with breast cancer positive for SSTR2.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess objective response in study participants receiving lutetium Lu 177 dotatate (177Lu-DOTATATE) therapy.

SECONDARY OBJECTIVES:

I. Assess the rate of disease control following 177Lu-DOTATATE therapy. II. Evaluate duration of treatment response to 177Lu-DOTATATE. III. Assess progression-free survival (PFS). IV. Assess safety and tolerability of the 177Lu-DOTATATE therapy. V. Evaluate over time the requirements for stable disease.

OUTLINE:

Patients receive 177Lu-DOTATATE intravenously (IV) over 30-40 minutes during weeks 1, 8, 16, and 24 in the absence of disease progression or unacceptable toxicity. Patients also receive gallium (Ga) 68-DOTATATE and undergo positron emission tomography/computed tomography (PET/CT) during screening, biopsy as clinically-indicated as well as CT and/or magnetic resonance imaging (MRI) and collection of blood samples throughout the study.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of > 6 months, as determined by the investigator
* Ability to understand and the willingness to sign a written informed consent document
* Patients aged >= 18-100 years old at time of informed consent
* Histologically or cytologically confirmed metastatic breast carcinoma
* Stage IV or recurrent disease with distant metastases
* Female and male patients with breast cancer will be included in the study
* Participants must have experienced disease progression after at least two lines of standard treatment modalities and/or one prior line of cytotoxic chemotherapy (not just endocrine therapy). Specifically, patients must have received or declined the following therapies: a) Hormone receptor positive (HR+)/HER2: endocrine therapy and CDK4/6 inhibitor (i); b) HER2+: trastuzumab, pertuzumab, T-DM1 and tucatinib; c) Triple negative breast cancer (TNBC): chemotherapy, immunotherapy (in PD-L1+ tumors). Patients can be consented if they are foregoing treatments known to confer survival advantage
* Participants must have at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v1).1 that is amendable to biopsy
* Confirmed presence of SSTR based on > 50% of lesions with DOTATATE uptake of 68Ga DOTATATE equivalent to the liver
* Participants must have fully recovered from the acute toxic effects of all prior treatment to grade 1 or less, except alopecia and =< grade 2 neuropathy which are allowed
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Participant must consent to undergo a pre-treatment screening biopsy for enrollment
* Hemoglobin >= 8.0 g/dL with no blood transfusion in the past 28 days (measured within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 2.0 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Platelet count >= 75 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Total bilirubin =< 3 x institutional upper limit of normal (ULN) (measured within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (unless liver metastases are present in which case they must be =< 5 x ULN) (measured within 28 days prior to administration of study treatment)
* Serum albumin >= 3.0 g/L, unless prothrombin time or international normalized ratio (INR) value is within the normal range (measured within 28 days prior to administration of study treatment)
* Participants must have serum creatinine =< 1.7 mg/dL, or creatinine clearance estimated of >= 51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test (measured within 28 days prior to administration of study treatment)
* Female participants of childbearing potential (FOCBP) must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* FOCBP agree to use a highly-effective method of contraception starting with the first dose of study therapy up to 7 months after the last dose of study therapy

  * FOCBP are those who are not proven postmenopausal. Postmenopausal is defined as:

    * Amenorrheic for > 24 consecutive months following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50 years of age
    * Radiation-induced oophorectomy with last menses > 1 year ago
    * Chemotherapy-induced menopause with > 1 year interval since last menses
    * Surgical sterilization (bilateral oophorectomy or hysterectomy or tubal ligation)

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of first dose of 177Lu- DOTATATE treatment

  * Individuals in the follow-up phase of a prior investigational study may participate as long as it has been 4 weeks since last dose of the previous investigational agent or device
* Prior external beam radiation therapy to more than 25% of the bone marrow
* Other malignancy unless curatively treated with no evidence of disease for >= 5 years except: adequately treated non-melanoma skin cancer or curatively treated in situ cancer of the cervix
* Known brain metastases, unless these metastases have been treated and stabilized
* Peptide receptor radionuclide therapy at any time prior to study enrollment
* Known hypersensitivity to somatostatin analogues or any component of the 68Ga- DOTATATE or 177Lu- DOTATATE formulations
* Patients with uncontrolled infection will not be enrolled until infection is treated per provider discretion
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure
* Uncontrolled diabetes mellitus as defined by a fasting blood glucose > 2x ULN
* Any patient receiving treatment with short-acting somatostatin analogs, which cannot be interrupted for both 24 hours before and after the administration of 177Lu, or any patient receiving treatment with long-acting release somatostatin analogs that cannot be interrupted for at least 4 weeks before the administration of 177Lu- DOTATATE
* Any surgery or radiofrequency ablation within 12 weeks prior to enrollment in the study; or prior radioembolization; chemoembolization; or external beam radiation therapy (EBRT) to > 25% of bone marrow, at any time
* Any chemotherapy or targeted therapy within 4 weeks prior to enrollment in the study
* Current spontaneous urinary incontinence making impossible the safe administration of the radioactive study agent
* Any psychiatric illness that prevents patient from informed consent process
* Any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol
* Participant is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 months post-therapy
  Using the intent to treat (ITT) set and the efficacy analysis set, each ORR will be reported as a point estimate along with a 2-sided 95% exact confidence interval (CI).

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 3 months post-therapy
  A point estimate and 2-sided 95% CI will be provided for the DCR, defined as the proportion of participants achieving a complete response (CR), partial response (PR), or stable disease (SD) (as assessed by the investigator per Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1).
Duration of response (DOR) | Up to 12 months post-therapy
  DOR will be estimated on responding participants and plotted with cumulative incidence functions: one curve for the first occurrence of recurrence, progression, or disease-related death and one curve for deaths in the absence of disease recurrence or progression.
Progression-free survival | Up to 12 months post-therapy
  PFS will be plotted using a Kaplan-Meier curve and reported with median survival and a 95% CI.
Incidence of adverse events (AEs) | Up to 3 months post-therapy
  The severity of the AE will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Study drug-related AEs are those assessed by investigator as definitely or probably related. Using the safety analysis set, the incidence of treatment emergent adverse events (TEAEs) and non-treatment-related AEs will be determined for study participants who receive at least one dose of lutetium Lu 177 dotatate (177Lu- DOTATATE). The point estimate and 95% CI will be reported for overall toxicities as well as for each major organ category.
Duration of stable disease | Up to 12 months post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rodney F Pommier, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States